CLINICAL TRIAL: NCT00453362
Title: Pilot Study of Changes in FDG- and FLT-PET Imaging in Patients With Non-Small Cell Lung Cancer Following Treatment With Erlotinib
Brief Title: A Study of Changes in FDG- and FLT-PET Imaging in Patients With Non-Small Cell Lung Cancer Following Treatment With Erlotinib
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI3926g; ML20773
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2011-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Tarceva; Positron emission technology; PET; Computerized tomography; CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18; alovudine; Erlotinib Hydrochloride

ARMS (1):
- Erlotinib (Experimental): Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  After 14 days and after 56 days of treatment with Erlotinib participants underwent FDG-PET and FLT-PET scans.
  Interventions: Other: 2-deoxy-2-[18F]fluoro-D-glucose (FDG); Other: 3'-deoxy-3'-[18F]fluorothymidine (FLT); Drug: erlotinib HCl

INTERVENTIONS:
Other: 2-deoxy-2-[18F]fluoro-D-glucose (FDG) — FDG prepared in sterile buffered solution for intravenous injection. Dosage was based on the participant's weight not to exceed 15 mCi (millicurie).
Other: 3'-deoxy-3'-[18F]fluorothymidine (FLT) — FLT 7 mCi dose prepared in sterile buffered solution for intravenous injection.
Drug: erlotinib HCl — Tablets taken orally 150 mg/day.
  Other Names: Tarceva

SUMMARY:
This is a single-arm, open-label, multicenter, international pilot study to evaluate changes that occur in 2-deoxy-2-[18F]fluoro-D-glucose (FDG)- and 3'-deoxy-3'-[18F]fluorothymidine(FLT)-PET (Positron Emission Tomography) imaging as a result of treatment with erlotinib in patients with recurrent or refractory non-small cell lung cancer (NSCLC). The study will enroll approximately 30 patients at approximately 4 sites in Australia and 2 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form(s)
* Histologically confirmed NSCLC
* Recurrent or progressive disease after receiving at least one chemotherapy regimen for advanced or metastatic NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Age ≥ 18 years
* Recovery from reversible acute effects of prior anti-cancer therapy (chemotherapy, radiotherapy, or investigational treatment) to NCI Common Toxicity Criteria for Adverse Events (NCI CTCAE) Grade ≤ 1 (excluding alopecia)
* Ability to comply with the study and follow-up procedures, including all specified imaging studies
* Ability to take oral medication
* Availability of archival diagnostic paraffin-embedded tumor tissue and willingness to provide sufficient tissue for testing for EGFR levels in tumor by both immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH)
* Life expectancy ≥ 3 months
* Measurable disease on computed tomography (CT)
* At least one detectable lesion on FDG-PET scan and/or FLT-PET scan that is measurable on CT
* Use of an acceptable means of contraception (men and women of childbearing potential) or documentation of infertility

Exclusion Criteria:

* Prior treatment with an investigational or marketed agent for the purpose of inhibiting epidermal growth factor receptor (EGFR) (including, but not limited to, erlotinib and gefitinib)
* Chemotherapy, radiotherapy, or investigational treatment within 14 days or within 5 half-lives of the active molecules in the chemotherapy or investigational treatment, whichever is longer, prior to study entry or from which patients have not yet recovered
* Inability to take oral medications, disease affecting gastrointestinal absorption, or prior surgical procedure affecting gastrointestinal absorption
* Uncontrolled diabetes
* Any unstable systemic disease (including active infection, unstable angina, congestive heart failure, myocardial infarction within 1 month prior to study entry, hepatic, renal, or metabolic disease)
* Pregnancy or lactation
* History of another malignancy in the past 2 years, unless the malignancy has been adequately treated, is currently not detectable, and is associated with a 5-year survival > 90%
* Claustrophobia
* Any other disease, condition, physical examination finding, or clinical laboratory finding which, in the opinion of the investigator, makes the patient inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fine, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single-arm, open-label, multicenter, international pilot study. The study was expected to enroll approximately 100 evaluable patients at approximately eight sites in Australia and the United States. The study was initiated on 6 DEC 2006 and completed on 23 APR 2010.
Groups:
- Erlotinib: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  After 14 days and after 56 days of treatment with Erlotinib participants underwent FDG-PET (2-deoxy-2-[18F]fluoro-D-glucose-Positron Emission Tomogrpahy)and FLT-PET (3'-deoxy-3'-[18F]fluorothymidine-Positron Emission Tomogrpahy) scans.
  FDG-PET intravenous injection dosage was based on participant's weight not to exceed 15 mCi and FLT-PET intravenous dose was 7 mCi.
Period: Overall Study
Arm/Group | Erlotinib
Started | 88 (14 participants consented but did not receive drug and are not represented in the baseline data)
Treated With Erlotinib | 74
FDG-PET Evaluable | 51 (Participants who completed all FDG-PET scans through day 56.)
FLT-PET Evaluable | 50 (Participants who completed all FLT-PET scans through day 56.)
Completed | 1
Not Completed | 87
Not completed — Adverse Event | 5
Not completed — Death | 7
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Progression of disease | 56
Not completed — Screening Failure | 14

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
Arm/Group | Erlotinib
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: years] — Patients who were treated with any dose of erlotinib were included in the summary of baseline measures.
  years | 62.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) of Groups by FDG Response at Day 56
Description: PFS was defined as the time from the date of first erlotinib dose to disease progression or death, whichever occurs first.
  PFS was compared between patients with FDG-PET response and patients without FDG-PET response, independent of CT response (per RECIST 1.0) at Day 56 of treatment with erlotinib.
  Mean of the percent changes in maximal standard uptake values (mSUVmax) from FDG-PET scans was used to define FDG-PET response. Based on European Organization for Research on the Treatment of Cancer (EORTC) definitions, an objective FDG-PET response was defined an mSUVmax <-25%.
Time Frame: Time from first erlotinib treatment to disease progression on CT (per RECIST 1.0) or death, whichever occurs first, assessed up to 2 years
Population: FDG-Evaluable Patients. Participants who were treated with erlotinib and underwent all FDG-PET scans through Day 56 were included in the analysis. Censoring occurred at the date of the last tumor assessment.
Measure: Median (Full Range); unit: weeks
Groups:
- Erlotinib_FDG Responders: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight not to exceed 15 mCi. Patients who had CR/PR on FDG-PET scans at Day 56 were included in this group.
- Erlotinib_ FDG Non-Responders: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight not to exceed 15 mCi. Patients who did not have CR/PR on FDG-PET scans at Day 56 were included in this group.
Arm/Group | Erlotinib_FDG Responders | Erlotinib_ FDG Non-Responders
Number analyzed (Participants) | 6 | 45
weeks | 28.1 [16.14 to 40.14] | 12.1 [7.86 to 51.14]
Statistical Analysis 1: Comparison: Erlotinib_FDG Responders vs Erlotinib_ FDG Non-Responders; The null hypothesis is that there is no difference in PFS between FDG Responders and FDG Non-Responders. The alternative hypothesis is that FDG Responders would have prolonged PFS compared with FDG Non-Responders; Test type: Superiority or Other; p = 0.017, Log Rank — This comparison is for hypothesis generation, rather than hypothesis testing. Thus the p-value is not adjusted for multiple comparisons, and the interpretation of p-value should be with caution; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.11 to 0.87] — The hazard ratio was estimated using a Cox Proportional Hazard Model. The hazard ratio is relative to FDG Non-Responders

2. Secondary Outcome: Percentage of Patients With FDG-PET Responses
Description: In patients with computed tomography (CT)-stable disease (according to RECIST 1.0) at 56 days of erlotinib treatment, the percentage of patients who demonstrated FDG-PET responses after the initial 14 days and 56 days of erlotinib treatment.
  FDG-PET response was defined as a mSUVmax from FDG-PET scans <-25%.
  CT SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: Day 14 and Day 56
Population: FDG-Evaluable patients. Participants who were treated with erlotinib, underwent all FDG-PET scans through Day 56 and had stable disease by CT at Day 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Erlotinib: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight not to exceed 15 mCi.
Arm/Group | Erlotinib
Number analyzed (Participants) | 26
Percentage of Participants
  Day 14 response | 7.7 [1.4 to 23.4]
  Day 56 response | 11.5 [3.2 to 29.9]

3. Primary Outcome: PFS of Patients With FDG-PET Complete Response (CR)/Partial Response (PR) Versus FDG-PET Progressive Disease (PD) in Patients With Computed Tomography (CT) Stable Disease (SD) at Day 56
Description: PFS was defined as the time from the date of first erlotinib dose to disease progression or death, whichever occurs first.
  PFS was compared between patients with FDG-PET response (Complete /Partial Responses) and patients with FDG-PET progression, within the subset of patients who demonstrated stable disease on CT (per RECIST 1.0) at Day 56 of treatment with erlotinib. FDG-PET response; defined as a mSUVmax from FDG-PET scans of <-25% and FDG-PET disease progression; defined as a mSUVmax >+25% or the development of a new lesion with a mSUVmax above background not explained by another cause.
Time Frame: as for outcome 1
Population: FDG-Evaluable patients were treated with erlotinib, underwent all FDG-PET scans through Day 56 and had SD by CT at Day 56. Censoring at last tumor assessment.
  CT SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since treatment start.
Measure: Median (Full Range); unit: weeks
Groups:
- Erlotinib_FDG Responders With CT SD at Day 56: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight not to exceed 15 mCi. Patients who had CR/PR on FDG-PET scans at Day 56 were included in this group.
- Erlotinib_FDG Progressive Disease With CT SD at Day 56: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight not to exceed 15 mCi. Patients who had Progressive disease on FDG-PET scans at Day 56 were included in this group.
Arm/Group | Erlotinib_FDG Responders With CT SD at Day 56 | Erlotinib_FDG Progressive Disease With CT SD at Day 56
Number analyzed (Participants) | 3 | 10
weeks | 32.1 [18 to 32.14] | 14.9 [8.14 to 32.14]
Statistical Analysis 1: Comparison: Erlotinib_FDG Responders With CT SD at Day 56 vs Erlotinib_FDG Progressive Disease With CT SD at Day 56; The null hypothesis is that there is no difference in PFS between FDG Responders and FDG Progressive Disease. The alternative hypothesis is that FDG Responders would have a prolonged PFS compared to FDG Progressive Disease; Test type: Superiority or Other; p = 0.076, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.06 to 1.42] — The hazard ratio was estimated using a Cox Proportional Hazard Model. The hazard ratio is relative to FDG Progressive Disease

4. Secondary Outcome: Percentage of Patients With FLT-PET Responses
Description: In patients with CT-stable disease (according to RECIST 1.0) at 56 days of erlotinib treatment, the percentage of patients who demonstrated FLT-PET responses after the initial 14 days and 56 days of erlotinib treatment.
  FLT-PET response was defined as a mSUVmax from FLT-PET scans <-25%. CT SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: Day 14 and Day 56
Population: FLT-Evaluable Patients. Participants who were treated with erlotinib, underwent all FLT-PET scans through Day 56 and had stable disease by CT at Day 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Erlotinib: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FLT-PET was scheduled on screening, Day 14 and Day 56. FLT intravenous injection dose was 7 mCi.
Arm/Group | Erlotinib
Number analyzed (Participants) | 26
Percentage of Participants
  Day 14 response | 7.7 [1.4 to 23.4]
  Day 56 response | 7.7 [1.4 to 23.4]

5. Primary Outcome: Progression Free Survival of Groups by FLT Response at Day 56
Description: PFS was defined as the time from the date of first erlotinib dose to disease progression or death, whichever occurs first.
  PFS was compared between patients with FLT-PET response and patients without FLT-PET response, independent of CT response (per RECIST 1.0) at Day 56 of treatment with erlotinib.
  FLT-PET response was defined as a mSUVmax from FLT-PET scans <-25%.
Time Frame: as for outcome 1
Population: FLT-Evaluable Patients. Participants who were treated with erlotinib and underwent all FLT-PET scans through Day 56 were included in the analysis. Censoring occurred at the date of the last tumor assessment.
Measure: Median (Full Range); unit: weeks
Groups:
- Erlotinib_FLT Responders: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FLT-PET was scheduled on screening, Day 14 and Day 56. FLT intravenous injection dose was 7 mCi. Patients who had CR/PR on FLT-PET scans at Day 56 were included in this group.
- Erlotinib_ FLT Non-Responders: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FLT-PET was scheduled on screening, Day 14 and Day 56. FLT intravenous injection dose was 7 mCi. Patients who did not have CR/PR on FLT-PET scans at Day 56 were included in this group.
Arm/Group | Erlotinib_FLT Responders | Erlotinib_ FLT Non-Responders
Number analyzed (Participants) | 4 | 46
weeks | 39.9 [18 to 40.14] | 13.1 [7.86 to 51.14]
Statistical Analysis 1: Comparison: Erlotinib_FLT Responders vs Erlotinib_ FLT Non-Responders; The null hypothesis is that there is no difference in PFS between FLT Responders and FLT Non-Responders. The alternative hypothesis is that FLT Responders would have prolonged PFS compared with FLT Non-Responders; Test type: Superiority or Other; p = 0.008, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.04 to 0.73] — The hazard ratio was estimated using a Cox Proportional Hazard Model. The hazard ratio is relative to FLT Non-Responders

6. Primary Outcome: Progression Free Survival of Patients With FLT CR/PR Versus FLT PD in Patients With CT SD at Day 56
Description: PFS was defined as the time from the date of first erlotinib dose to disease progression or death, whichever occurs first.
  PFS was compared between patients with FLT-PET response and patients without FLT-PET response, independent of computed tomography (CT) response (per RECIST 1.0) at Day 56 of treatment with erlotinib.
  FLT-PET response was defined as a mSUVmax from FLT-PET scans <-25% and FLT-PET disease progression was defined as a mSUVmax from FLT-PET scans >+25% or the development of a new lesion with a mSUVmax above background not explained by another cause.
Time Frame: as for outcome 1
Population: FLT-Evaluable patients were treated with erlotinib, underwent all FLT-PET scans through Day 56 and had SD by CT at Day 56. Censoring at last tumor assessment.
  CT SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since treatment start.
Measure: Median (Full Range); unit: weeks
Groups:
- Erlotinib_FLT Responders With CT SD at Day 56: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FLT-PET was scheduled on screening, Day 14 and Day 56. FLT intravenous injection dose was 7 mCi. Patients who had CR/PR on FLT-PET scans at Day 56 were included in this group.
- Erlotinib_FLT Progressive Disease With CT SD at Day 56: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FLT-PET was scheduled on screening, Day 14 and Day 56. FLT intravenous injection dose was 7 mCi. Patients who had Progressive disease on FLT-PET scans at Day 56 were included in this group.
Arm/Group | Erlotinib_FLT Responders With CT SD at Day 56 | Erlotinib_FLT Progressive Disease With CT SD at Day 56
Number analyzed (Participants) | 2 | 4
weeks | NA [18 to 24] — Not applicable. The median PFS of Day 56 FLT-PET responders was not estimable using Kaplan-Meier methodology. Hazard ratio and confidence interval are not estimable due to the limited number of events. | 12.9 [8.29 to 17.29]
Statistical Analysis 1: Comparison: Erlotinib_FLT Responders With CT SD at Day 56 vs Erlotinib_FLT Progressive Disease With CT SD at Day 56; The null hypothesis is that there is no difference between FLT Responders and FLT Progressive Disease. Alternative hypothesis is that FLT responders would have prolonged PFS compared to FLT Progressive Disease; Test type: Superiority or Other; p = 0.049, Log Rank — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Overall Survival of Groups by FDG Response at Day 56
Description: Overall survival (OS) was defined as the time from the date of first erlotinib dose to death.
  Overall survival (OS) was compared between patients with FDG-PET response and patients without FDG-PET response, independent of Response Evaluation Criteria in Solid Tumors (RECIST 1.0) computed tomography (CT) response at Day 56 of treatment with erlotinib. FDG-PET response was defined as a mSUVmax from FDG-PET scans <-25%.
Time Frame: From first erlotinib treatment to death, assessed up to 2 years
Population: FDG-Evaluable Patients. Participants who were treated with erlotinib and underwent all FDG-PET scans through Day 56 were included in the analysis. Censoring occurred at the last date patients known to be alive.
Measure: Median (Full Range); unit: months
Groups:
- Erlotinib_ FDG Non-Responder: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight not to exceed 15 mCi. Patients who did not have CR/PR on FDG-PET scans at Day 56 were included in this group.
Arm/Group | Erlotinib_FDG Responders | Erlotinib_ FDG Non-Responder
Number analyzed (Participants) | 6 | 45
months | NA [4.99 to 23.98] — Not applicable. The median OS of Day 56 FDG-PET responders was not estimable using Kaplan-Meier methodology. | 7.8 [1.94 to 24.51]
Statistical Analysis 1: Comparison: Erlotinib_FDG Responders vs Erlotinib_ FDG Non-Responder; The null hypothesis is that there is no difference in OS between FDG Responders and FDG Non-Responders. The alternative hypothesis is that FDG responders would have prolonged OS compared with FDG Non-Responders; Test type: Superiority or Other; p = 0.073, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.11 to 1.16] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: FDG Response in Subgroups by CT Response at Day 56
Description: In patients with partial response or progressive disease on CT (per RECIST 1.0) after 56 days of erlotinib treatment, the percentage of patients who demonstrated FDG-PET responses on Day 56 defined as a mSUVmax from FDG-PET scans <-25%.
  CT Partial Response defined as a 30% decrease in the sum of the longest diameter (LD) of target lesion taking as reference the baseline sum of the LD.
  CT Progressive disease defined as a 20% increase in the sum of the longest diameter of target lesions taking as reference the smallest sum LD since treatment started or appearance of 1 or more new lesions.
Time Frame: Day 56
Population: FDG-Evaluable Patients. Participants who were treated with erlotinib and underwent all FDG-PET scans through Day 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Erlotinib: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  FDG-PET was scheduled on screening, Day 14 and Day 56. FDG intravenous injection-dosage based on participant's weight no to exceed 15 mCi.
Arm/Group | Erlotinib
Number analyzed (Participants) | 51
Percentage of participants
  CT Partial response (n=4) | 75 [24.9 to 98.7]
  CT Progressive Disease (n=21) | 0 [0 to 14.6]

9. Secondary Outcome: FLT Response in Subgroups by CT Response at Day 56
Description: In patients with partial response or progressive disease on CT (per RECIST 1.0) after 56 days of erlotinib treatment, the percentage of patients who demonstrated FLT-PET responses on Day 56 defined as a mSUVmax from FLT-PET scans <-25%.
  CT Partial Response defined as a 30% decrease in the sum of the longest diameter (LD) of target lesion taking as reference the baseline sum of the LD.
  CT Progressive disease defined as a 20% increase in the sum of the longest diameter of target lesions taking as reference the smallest sum LD since treatment started or appearance of 1 or more new lesions.
Time Frame: Day 56
Population: FLT-Evaluable Patients. Participants who were treated with erlotinib and underwent all FLT-PET scans through Day 56 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 50
Percentage of participants
  CT Partial response (n=4) | 50 [9.8 to 90.2]
  CT Progressive Disease (n=20) | 0 [0 to 15.4]

10. Primary Outcome: Overall Survival of Patients With FDG CR/PR Versus FDG PD in Patients With CT SD at Day 56
Description: Overall survival (OS) was defined as the time from the date of first erlotinib dose to death.
  OS was compared between patients with FDG-PET response and patients with FDG-PET progression, within the subset of patients who demonstrated stable disease (SD) on CT (per RECIST 1.0) at Day 56 of treatment with erlotinib.
  FDG-PET response was defined as a mSUVmax from FDG-PET scans <-25% and FDG-PET disease progression was defined as a mSUVmax from FDG-PET scans >+25% or the development of a new lesion with a mSUVmax above background not explained by another cause.
Time Frame: From first erlotinib treatment to death, assessed up to 2 years
Population: Patients who were treated with erlotinib, underwent all FDG-PET scans thru Day 56 and had SD by CT at Day 56. Censoring at last date patients known to be alive.
  CT SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since treatment start.
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib_FDG Responders With CT SD at Day 56 | Erlotinib_FDG Progressive Disease With CT SD at Day 56
Number analyzed (Participants) | 3 | 10
months | 12.2 [4.99 to 17.84] | 8.8 [2.37 to 20.07]
Statistical Analysis 1: Comparison: Erlotinib_FDG Responders With CT SD at Day 56 vs Erlotinib_FDG Progressive Disease With CT SD at Day 56; The null hypothesis is that there is no difference in Overall Survival between FDG Responders and FDG Progressive Disease. The alternative hypothesis is that FDG Responders would have prolonged OS compared with FDG Progressive Disease; Test type: Superiority or Other; p = 0.618, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.14 to 3.21] — [estimate comment as in outcome 3, analysis 1]

11. Primary Outcome: Overall Survival of Groups by FLT Response at Day 56
Description: Overall survival (OS) was defined as the time from the date of first erlotinib dose to death.
  OS was compared between patients with FLT-PET response and patients without FLT-PET response, independent of CT response (per RECIST 1.0) at Day 56 of treatment with erlotinib.
  FLT-PET response was defined as a mSUVmax from FLT-PET scans <-25%.
Time Frame: From first erlotinib treatment to death, assessed up to 2 years
Population: FLT-Evaluable Patients. Participants who were treated with erlotinib and underwent all FLT-PET scans through Day 56 were included in the analysis. Censoring occurred at the last date patients known to be alive.
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib_FLT Responders | Erlotinib_ FLT Non-Responders
Number analyzed (Participants) | 4 | 46
months | NA [4.99 to 23.98] — Not applicable. The median OS of Day 56 FLT-PET responders was not estimable using Kaplan-Meier methodology. | 8.4 [1.94 to 24.51]
Statistical Analysis 1: Comparison: Erlotinib_FLT Responders vs Erlotinib_ FLT Non-Responders; The null hypothesis is that there is no difference in OS between FLT Responders and FLT Non-Responders. The alternative hypothesis is that FLT Responders would have prolonged OS compared with FLT Non-Responders; Test type: Superiority or Other; p = 0.163, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.09 to 1.57] — [estimate comment as in outcome 5, analysis 1]

12. Primary Outcome: Overall Survival of Patients With FLT CR/PR Versus FLT PD in Patients With CT SD at Day 56
Description: Overall survival (OS) was defined as the time from the date of first erlotinib dose to death.
  OS was compared between patients with FLT-PET response and patients with FLT-PET progression, within the subset of patients who demonstrated SD on CT (per RECIST 1.0) at Day 56 of treatment with erlotinib.
  FLT-PET response was defined as a mSUVmax from FLT-PET scans of <-25% and FLT-PET disease progression was defined as a mSUVmax from FLT-PET scans >+25% or the development of a new lesion with a mSUVmax above background not explained by another cause.
Time Frame: From first erlotinib treatment to death, assessed up to 2 years
Population: Patients who were treated with erlotinib,underwent all FLT-PET scans thru Day 56 and had SD by CT at Day 56. Censoring at last date patients known to be alive.
  CT SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started.
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib_FLT Responders With CT SD at Day 56 | Erlotinib_FLT Progressive Disease With CT SD at Day 56
Number analyzed (Participants) | 2 | 4
months | NA [4.99 to 17.84] — Not applicable. The median OS of Day 56 FLT-PET responders was not estimable using Kaplan-Meier methodology. | 8 [2.37 to 14.29]
Statistical Analysis 1: Comparison: Erlotinib_FLT Responders With CT SD at Day 56 vs Erlotinib_FLT Progressive Disease With CT SD at Day 56; The null hypothesis is that there is no difference in OS between FLT Responders and FLT Progressive Disease. The alternative hypothesis is that FLT Responders would have prolonged OS compared with FLT Progressive Disease; Test type: Superiority or Other; p = 0.327, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.04 to 3.16] — The hazard ratio was estimated using a Cox Proportional Hazard Model. The hazard ratio is relative to FLT Progressive Disease

13. Secondary Outcome: Number of Participants With Adverse Events Due to FLT-PET Imaging
Description: The number of participants who experienced an adverse event judged by the investigator to be related to FLT-PET.
Time Frame: From screening to Day 112 assessment visit or study discontinuation or termination, whichever is first. On visits after Day 112, only SAE were recorded.
Population: Patients with non-small cell lung cancer (NSCLC) who underwent FLT-PET scans.
Measure: Number; unit: Participants
Groups:
- Overall Study Participants: All Participants who underwent any FLT-PET scan during the study (including screening) were included in the analysis.
  FLT-PET was scheduled on screening, Day 14 and Day 56. FLT intravenous injection dose was 7 mCi.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 85
Participants | 0

ADVERSE EVENTS:
Time Frame: Screening to Day 112 assessment visit or study discontinuation or termination, whichever is earlier. On visits after Day 112, only Serious Adverse Events were recorded. (Up to 1 year)
Description: Includes evaluation of all Safety-Evaluable Patients [n = 85].
Groups:
- Erlotinib: Erlotinib 150 mg/day taken orally at approximately the same time of day with 200 mL (6-8 Ounces) of water on an empty stomach. Participants received Erlotinib for 1 year or until they developed progressive disease or intolerable toxicity.
  After 14 days and after 56 days of treatment with Erlotinib, participants underwent FDG-PET and FLT-PET scans. FDG-PET intravenous injection-dosage based on participant's weight not to exceed 15 mCi and FLT-PET intravenous dose of 7 mCi.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 37/85
Other Adverse Events (participants affected / at risk) | 46/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=85)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
DISEASE PROGRESSION (General disorders) | 5
FATIGUE (General disorders) | 2
PYREXIA (General disorders) | 2
PNEUMONIA (Infections and infestations) | 4
BRONCHITIS (Infections and infestations) | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1
GANGRENE (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1
FALL (Injury, poisoning and procedural complications) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEADACHE (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
PRESYNCOPE (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 3
DEPRESSION (Psychiatric disorders) | 1
DISORIENTATION (Psychiatric disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=85)
ANAEMIA (Blood and lymphatic system disorders) | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
MELAENA (Gastrointestinal disorders) | 1
FATIGUE (General disorders) | 6
DISEASE PROGRESSION (General disorders) | 5
PAIN (General disorders) | 2
PYREXIA (General disorders) | 1
PNEUMONIA (Infections and infestations) | 4
BRONCHITIS (Infections and infestations) | 1
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
DERMATITIS INFECTED (Infections and infestations) | 1
GANGRENE (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
PARONYCHIA (Infections and infestations) | 1
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1
BLOOD GLUCOSE INCREASED (Investigations) | 2
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
HEADACHE (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
NEURALGIA (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
SCIATICA (Nervous system disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 2
ANXIETY (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
DISORIENTATION (Psychiatric disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 5
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1
HYPOTENSION (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.